CLINICAL TRIAL: NCT02729974
Title: Use of ROTEM Intraoperatively in Women With Placenta Accreta
Acronym: ROTEM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Heather Campbell, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 81113
Record Dates: First submitted 2016-03-18; First posted 2016-04-06 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Placenta Accreta
Keywords: thromboelastography
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ROTEM (Experimental): Participants randomized to this arm will have rapid testing of hematocrit and clotting function every 30 minutes during the hysterectomy portion of their surgery for placenta accreta, with transfusion of blood products based on defined abnormalities in these tests.
  Interventions: Procedure: ROTEM
- Standard treatment (Active Comparator): Participants randomized to this arm will have standard visual assessment of blood loss and standard laboratory studies to assess blood count and clotting function when indicated during the hysterectomy portion of their surgery for placenta accreta. Transfusion of blood products will be based on abnormalities of these test results.
  Interventions: Procedure: standard treatment

INTERVENTIONS:
Procedure: ROTEM — rapid testing of blood clot formation
  Arms: ROTEM
Procedure: standard treatment — visual assessment of blood loss and clotting function every 30 minutes, combined with standard laboratory testing when indicated
  Arms: Standard treatment

SUMMARY:
This study evaluates the use of rapid tests for hematocrit and clotting function in women undergoing surgery for placenta accreta. Half of participants will have these rapid tests performed during surgery to guide blood product transfusion and the other half will have standard lab tests performed to guide transfusion.

DETAILED DESCRIPTION:
Placenta accreta has become an increasingly common pregnancy complication. Serious complications are common in patients with placenta accreta, including hemorrhage, transfusion of blood products, abdominal organ injury, bladder surgery, and ICU admission. Hemorrhage, or excessive blood loss, is the most common complication and often results in impaired ability for the body to form blood clots normally.

The development of rapid testing of hematocrit and clotting function may allow for earlier identification of patients who have severe blood loss and development of clotting abnormalities. The investigators are testing whether use of this technology in patients undergoing surgery for placenta accreta, with earlier identification of patients with severe blood loss or clotting abnormality, will result in a lower need for transfusion and fewer complications.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with placenta accreta during pregnancy who are scheduled to have delivery by cesarean section with hysterectomy to follow.

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of units of blood products transfused | From the time of surgery up to 10 days, or until discharge from the hospital if this occurs earlier

SECONDARY OUTCOMES:
Number of hours spent in ICU | From the time of surgery up to 10 days, or until discharge from the hospital if this occurs earlier
Number of days in the hospital | From the time of surgery up to 10 days, or until discharge from the hospital if this occurs earlier
Presence of infection at the surgery site | From the time of surgery up to 10 days, or until discharge from the hospital if this occurs earlier
Readmission for other complications | For up to 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heather Campbell, MD, Principal Investigator — University of Utah, Department of OBGYN

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wortman AC, Alexander JM. Placenta accreta, increta, and percreta. Obstet Gynecol Clin North Am. 2013 Mar;40(1):137-54. doi: 10.1016/j.ogc.2012.12.002. PMID 23466142
- [Background] Upson K, Silver RM, Greene R, Lutomski J, Holt VL. Placenta accreta and maternal morbidity in the Republic of Ireland, 2005-2010. J Matern Fetal Neonatal Med. 2014 Jan;27(1):24-9. doi: 10.3109/14767058.2013.799654. Epub 2013 May 30. PMID 23638753
- [Background] Eller AG, Bennett MA, Sharshiner M, Masheter C, Soisson AP, Dodson M, Silver RM. Maternal morbidity in cases of placenta accreta managed by a multidisciplinary care team compared with standard obstetric care. Obstet Gynecol. 2011 Feb;117(2 Pt 1):331-337. doi: 10.1097/AOG.0b013e3182051db2. PMID 21309195
- [Background] Meyer AS, Meyer MA, Sorensen AM, Rasmussen LS, Hansen MB, Holcomb JB, Cotton BA, Wade CE, Ostrowski SR, Johansson PI. Thrombelastography and rotational thromboelastometry early amplitudes in 182 trauma patients with clinical suspicion of severe injury. J Trauma Acute Care Surg. 2014 Mar;76(3):682-90. doi: 10.1097/TA.0000000000000134. PMID 24553534
- [Background] Brazzel C. Thromboelastography-guided transfusion Therapy in the trauma patient. AANA J. 2013 Apr;81(2):127-32. PMID 23971232
- [Background] Rourke C, Curry N, Khan S, Taylor R, Raza I, Davenport R, Stanworth S, Brohi K. Fibrinogen levels during trauma hemorrhage, response to replacement therapy, and association with patient outcomes. J Thromb Haemost. 2012 Jul;10(7):1342-51. doi: 10.1111/j.1538-7836.2012.04752.x. PMID 22519961
- [Background] Huissoud C, Carrabin N, Audibert F, Levrat A, Massignon D, Berland M, Rudigoz RC. Bedside assessment of fibrinogen level in postpartum haemorrhage by thrombelastometry. BJOG. 2009 Jul;116(8):1097-102. doi: 10.1111/j.1471-0528.2009.02187.x. Epub 2009 May 12. PMID 19459866